CLINICAL TRIAL: NCT00628134
Title: Self-dispersing Liquids as Aerosol Drug Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Tim Corcoran, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO07090095; CORCOR07A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation Therapeutics)
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; surfactant; aerosol; inhaled drug; inhaled antibiotic
MeSH Terms: conditions — Cystic Fibrosis | interventions — calfactant; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects inhaled calfactant then isotonic saline
  Interventions: Drug: calfactant; Drug: isotonic saline
- 2 (Experimental): Subjects inhaled isotonic saline then calfactant
  Interventions: Drug: calfactant; Drug: isotonic saline

INTERVENTIONS:
Drug: calfactant — single inhaled dose by nebulizer
  Other Names: Infasurf
Drug: isotonic saline — single inhaled dose by nebulizer

SUMMARY:
Inhaled medications are often used to treat lung diseases such as cystic fibrosis. We are performing this study to determine whether inhaled medications dissolved in surfactant-based solutions will distribute more evenly throughout the lungs when compared to standard saline-based solutions. We think that inhaling medication that is in a surfactant-based liquid will result in more medication reaching partially blocked parts of the lung. This study will use a special nuclear medicine test called an aerosol deposition scan to compare how a drug spreads in the lung using a surfactant-based aerosol compared to a saline-based aerosol.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an inherited chronic disease that affects the lungs and digestive system of about 30,000 children and adults in the United States (70,000 worldwide). The lungs of a person with cystic fibrosis often contain thick sticky mucus that can clog the lungs and lead to life-threatening lung infections. A major milestone in the treatment of CF was the development of an inhaled form of an antibiotic drug called tobramycin. For an inhaled antibiotic to work it must be delivered to all infected parts of the lung. Many studies have shown that blockages in the lungs, like those found in CF patients, can prevent inhaled medicines from reaching all parts of the lungs.

Usually aerosolized medications are dissolved in saline or water. Most of these medications could be dissolved in surfactant solutions and aerosolized. Soaps are common examples of surfactants. Surfactants may have the ability to spread medication over the inside surface of the lungs similar to the way dish soap spreads over water. We think that inhaling medication that is in a surfactant-based liquid will result in more medication reaching partially blocked parts of the lung. We further believe that the normal movements of the lung associated with breathing will further spread surfactant-based aerosol medications, and contribute to even more even drug distribution over longer periods of time.

A surfactant-based inhaled antibiotic would have the potential to reach more sites of infection in the lung, possibly getting rid of infection all together. This study will use a special test called an aerosol deposition scan to compare how a drug spreads in the lung using a surfactant-based aerosol compared to a saline-based aerosol. The study includes one screening and two testing visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms
* Clinically stable as determined by the investigator (pulmonologist).

Exclusion Criteria:

* Known allergies to any of the administered components (as described by subjects or based on positive RAST test to bovine serum albumin)
* Any past instances of bronchospasm associated with aerosol medications
* FEV1 < 60% predicted
* Positive urine pregnancy test (as administered to all female subjects of childbearing potential on testing days)
* Currently a nursing mother
* History of reactive airways disease associated with significant instances of bronchoconstriction
* Self-reported smoking history within the last 6 months.
* Subjects receiving any treatments or diagnostic procedures involving radioisotopes within the last 30 days.
* Subjects in the CF arm of the study will also be excluded if their pre-study pulmonary function test (FEV1) is more than 15% depressed from their last baseline pulmonary function test, if this baseline value is from within the last 6 months, or if they have experienced an exacerbation requiring hospitalization or treatment with an IV antibiotic within the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Corcoran TE, Thomas KM, Garoff S, Tilton RD, Przybycien TM, Pilewski JM. Imaging the postdeposition dispersion of an inhaled surfactant aerosol. J Aerosol Med Pulm Drug Deliv. 2012 Oct;25(5):290-6. doi: 10.1089/jamp.2011.0920. Epub 2012 Mar 6. PMID 22393908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight subjects with cystic fibrosis were recruited.
Pre-assignment Details: Subjects performed two imaging study days. On one study day subjects inhaled Tc-SC particles suspended in calfactant. On the other study day they inhaled the same particles in saline. The order of the study days was randomized.
Groups:
- Surfactant Aerosol Then Saline Aerosol: cystic fibrosis patients who inhaled surfactant aerosol at the first study visit and saline aerosol at the second study visit
- Saline Aerosol Then Surfactant Aerosol: cystic fibrosis patients who inhaled saline aerosol at the first study visit and surfactant aerosol at the second study visit
Period: Overall Study
Arm/Group | Surfactant Aerosol Then Saline Aerosol | Saline Aerosol Then Surfactant Aerosol
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cystic fibrosis subjects
Groups:
- Cystic Fibrosis Subjects: Subjects with cystic fibrosis
  isotonic saline aerosol : single inhaled dose, 3ml by nebulizer
  calfactant aerosol : single inhaled dose, 3ml by nebulizer
Arm/Group | Cystic Fibrosis Subjects
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Uniformity of Aerosol Distribution
Description: Measured change in central/peripheral (c/p) dose ratio over a 30 minute period after aersol delivery (c/p at t=30 - c/p at t=0). Central and peripheral lung doses are measured as radioactive counts depicted on nuclear medicine gamma camera images after radioisotope aerosol delivery. The central lung zone is a rectangle with 1/2 the height and 1/2 the width of a box outlining the whole right lung. The peripheral lung zone is defined as the portion of the lung outside of the central lung zone. A change in c/p ratio over time would indicate transport of material from one lung zone to the other. The variable represents the realtive proportion of airways dosing to alveolar dosing - an indication of deposition uniformity in the lungs.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Subjects Inhaling Saline; Subjects Inhaling Surfactant: Subjects with cystic fibrosis
Arm/Group | Subjects Inhaling Saline | Subjects Inhaling Surfactant
Number analyzed (Participants) | 8 | 8
ratio | -0.05 (0.16) | 0.10 (0.10)
Statistical Analysis 1: Comparison: Subjects Inhaling Saline vs Subjects Inhaling Surfactant; Wilcoxon matched-pairs signed-ranks test was used for comparisons; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Peripheral Lung Dose
Description: Change over 30 minutes in the percentage of the total deposited aerosol dose found in the peripheral lung zone. We are reporting the %peripheral dose at t=30 minus the %peripheral dose at t=0. This dose is determined based on measured radioactive counts after aerosol delivery, using nuclear medicine gamma camera images. The central lung zone is defined as a rectangle with 1/2 the height and 1/2 the width of a rectangle that surrounds the right whole lung. The peripheral zone is the portion of the lung image not included in the central lung zone.
Time Frame: 30 minutes after delivery
Measure: Mean (Standard Deviation); unit: percentage of lung dose
Arm/Group | Subjects Inhaling Saline | Subjects Inhaling Surfactant
Number analyzed (Participants) | 8 | 8
percentage of lung dose | -3 (5) | -8 (8)
Statistical Analysis 1: Comparison: Subjects Inhaling Saline vs Subjects Inhaling Surfactant; Wilcoxon matched-pairs signed-ranks test was used for comparisons; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Subjects Inhaling Saline | Subjects Inhaling Surfactant
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Our aerosol delivery method resulted in more peripheral distribution than was anticipated. The more peripheral deposition pattern likely affected the location and quantity of deposited calfactant available to cause transport.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No